CLINICAL TRIAL: NCT00155753
Title: Genomewide Screening of Pathological Myopia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yung-Feng Shih, National Taiwan University Hospital
Other Study IDs: 9100205245
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-04

CONDITIONS: Pathological Myopia
Keywords: pathological myopia, genomic
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — DNA extracted from blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the possible candidate gene of pathological myopia

DETAILED DESCRIPTION:
High myopia (pathological myopia) is caused by excessive axial elongation that primarily involves the ora-equatorial area and the posterior pole. Peripheral fundus changes and posterior staphyloma formation are ophthalmoscopic evidences of this process. Pathological myopia often accompanied by glaucoma, cataracts, macular degeneration, and retinal detachment, leading to blindness when the damage to the retina is extremely severe. Population and family studies in Chinese have provided evidence for a genetic component to pathologic myopia. Children of myopic parents are more likely to have myopia than are children of nonmyopic parents. The ocular components (axial length, anterior chamber depth, and corneal curvature) and refractive errors of MZ twins are more closely aligned than are those of DZ twins.

Therefore, it is possible to search a potential candidate gene for myopia through the genomic study of pathological myopia.

ELIGIBILITY:
Inclusion Criteria:

* They are unrelated Chinese subjects with high myopia ≦-6.00D. The diagnosis of myopia is determined by the refractive error. Anisometropic individuals, with a refractive error of ≦-6.00 D for one eye and ≦-6.00 D for the other eye, with at least a 2-D difference between the two eyes, are considered unaffected.

Exclusion Criteria:

* Individuals are excluded if there is known ocular disease or insult that could predispose to myopia, such as retinopathy of prematurity or early-age media opacification, or if they had a known genetic disease associated with myopia, such as Stickler or Marfan syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Taiwanese
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2002-08; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Feng Shih, MD, Principal Investigator — National Taiwan University Hospiyal
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan